CLINICAL TRIAL: NCT02112487
Title: An Extension of AC-055-310, a Multi-center, Open-label, Single-arm, Phase 3b Study of Macitentan in Patients With Pulmonary Arterial Hypertension to Psychometrically Validate the French, Italian and Spanish Versions of the PAH-SYMPACT™
Brief Title: Extension of the Psychometric Validation Study ORCHESTRA in Patients With PAH
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Actelion (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AC-055-311
Record Dates: First submitted 2014-04-08; First posted 2014-04-14 (Estimated); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: pulmonary arterial hypertension; PAH-SYMPACT; PAH; psychometric instrument
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — macitentan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Macitentan (Experimental): 10 mg once daily
  Interventions: Drug: Macitentan

INTERVENTIONS:
Drug: Macitentan — 10 mg once daily
  Other Names: ACT-064992

SUMMARY:
Prospective, multi-center, open-label, single-arm, Phase 3b extension study of macitentan in patients with PAH.

To assess the long-term safety of macitentan in patients with pulmonary arterial hypertension (PAH) beyond treatment in the AC-055-310 study.

DETAILED DESCRIPTION:
To assess the long-term safety of macitentan in patients with pulmonary arterial hypertension (PAH) beyond treatment in the AC-055-310 study.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent prior to any study-mandated procedure.
2. Patients with PAH who completed the ORCHESTRA study (AC-055-310) as scheduled
3. Women of childbearing potential (as defined below) must:

   * Have a negative serum pregnancy test at Visit 1 (i.e., Visit 4 of study AC 055 310) and agree to perform monthly serum pregnancy tests.
   * Agree to use two reliable methods of contraception in parallel, from Visit 1 until 1 month after study drug discontinuation (see details below).

     * A female is considered to have childbearing potential unless she meets at least one of the following criteria:

       * Previous bilateral salpingo and/or oophorectomy, or hysterectomy.
       * Premature ovarian failure confirmed by a specialist.
       * Pre-pubescence, XY genotype, Turner syndrome, uterine agenesis.
       * Postmenopausal, defined as 12 consecutive months with no menses without an alternative medical cause.
     * Of the two contraceptive methods that must be used, one must be from Group 1, and one must be from Group 2, defined as follows:

       * Group 1: Oral, implantable, transdermal or injectable hormonal contraceptives, intrauterine devices, female sterilization (tubal ligation or non-surgical sterilization, e.g., permanent contraception with Essure procedure), or partner's sterilization (vasectomy). If a hormonal contraceptive is chosen from this group, it must be taken for at least one month prior to enrollment. Alternatively, if the Essure procedure is chosen as a contraceptive method, a hysterosalpingogram must have been performed to confirm correct location of the microinserts and tubal occlusion (as per manufacturer's recommendations).
       * Group 2: Female or male condoms, diaphragm or cervical cap, any of them in combination with a spermicide.
     * Sexual abstinence, rhythm methods, or contraception by the partner alone are not considered as acceptable methods of contraception for this study.

Exclusion Criteria:

1. Patients who prematurely discontinued study drug in study AC-055-310.
2. Females who are lactating or pregnant (positive Visit 1 pregnancy test) or plan to become pregnant during the study.
3. AST and/or ALT more than 3 X ULN.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2014-06-23 (Actual); Primary Completion 2018-09-19 (Actual); Study Completion 2018-09-19 (Actual)

PRIMARY OUTCOMES:
To assess the long-term safety of macitentan in patients with pulmonary arterial hypertension (PAH) beyond treatment in the AC-055-310 study. | Baseline to end of treatment visit (around 6 months on average)
  * Treatment-emergent adverse events (AEs)
  * AEs leading to premature discontinuation of study drug
  * Treatment-emergent serious adverse events (SAEs)
  * Proportion of patients with treatment-emergent ALT and/or AST abnormality (> 3, > 5, and > 8 x ULN) associated or not with total bilirubin > 2 x ULN.
  * Proportion of patients with treatment-emergent hemoglobin abnormality (≦ 100 g/L, and ≦ 80 g/L)

CONTACTS AND LOCATIONS:
Overall Officials: Loïc Perchenet, Study Director — Actelion
Locations (32):
- France (13):
  - Hôpital Louis Pradel, Bron
  - Hôpital Côte de Nacre, Caen
  - Hôpital Albert Michallon, Grenoble
  - CHU de Bicêtre, Le Kremlin-Bicêtre
  - CHRU Lille - Hôpital Cardiologique, Lille
  - Hôpital Arnaud de Villeneuve, Montpellier
  - Hôpitaux de Brabois, Nancy
  - Hôpital de Haut Levêque, Pessac
  - Hôpital Pontchaillou, Rennes
  - Hôpital Charles Nicolle, Rouen
  - Hôpital Nord, Saint-Etienne
  - Hôpital Civil, Strasbourg
  - Hôpital Larrey, Toulouse
- Italy (5):
  - Ospedale Sant'Orsola, Bologna
  - A.O.U.C. Careggi, Florence
  - UOC Immunologia Clinica B-PGRM Centro di Riferimento per la Sclerosi Sistemica, Rome
  - Centro Per La Diagnosi E La Cura Dell'Ipertensione Polmonare, Rome
  - Policlinico G.B. Rossi, Verona
- Spain (14):
  - Hospital General de Alicante, Alicante
  - Hospital Val Hebron, Barcelona
  - Hospital Clinic, Barcelona
  - Hospital de Cruces, Bilbao
  - Hospital Reina Sofia, Córdoba
  - Hospital Dr Negrin, Las Palmas de Gran Canaria
  - Hospital Universitario Insular Gran Canarias, Las Palmas de Gran Canaria
  - Hospital 12 Octubre, Madrid
  - Hospital La Paz, Madrid
  - Hospital Carlos Haya, Málaga
  - Hospital Son Espases, Palma de Mallorca
  - Hospital de Valdecilla, Santander
  - Hospital Virgen del Rocio, Seville
  - Hospita General U. Valencia, Valencia

REFERENCES:
- See also: Extension of the psychometric validation study ORCHESTRA in patients with PAH — http://www.clinicaltrialsregister.eu/ctr-search/trial/2013-003489-15/results